CLINICAL TRIAL: NCT03763019
Title: Correlation of Pulmonary Function Test and Ultrasonographic Diaphragm Measurements in Patients With Hemiplegia and Investigation of the Effects of Respiratory Exercises on These Parameters
Brief Title: Effects of Respiratory Exercises in Patients With Hemiplegia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bezmialem Vakif University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: 54022451-050.05.04
Record Dates: First submitted 2018-11-30; First posted 2018-12-04 (Actual); Last update posted 2020-02-05 (Actual); Status verified 2020-02

CONDITIONS: Hemiplegia; Respiratory Abnormality
Keywords: hemiplegia; respiratory function tests; respiratory exercises; diaphragm ultrasonography
MeSH Terms: conditions — Hemiplegia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Respiratory rehabilitation (Active Comparator): Conventional rehabilitation program aiming to normalize movement patterns and minimize spasticity. Including static and dynamic control of position, balance skills, weight shift, and activities of daily living. 45 minutes, once daily.
  Respiratory exercises 30 minutes, once daily, (incentive spirometric trainer, forced expiration, percussion, postural drainage etc.)
  Interventions: Procedure: Conventional rehabilitation; Procedure: Respiratory rehabilitation
- Conventional rehabilitation (Placebo Comparator): Conventional rehabilitation program aiming to normalize movement patterns and minimize spasticity. Including static and dynamic control of position, balance skills, weight shift, and activities of daily living. 45 minutes, once daily.
  Interventions: Procedure: Conventional rehabilitation

INTERVENTIONS:
Procedure: Conventional rehabilitation — Static and dynamic control of position, balance skills, weight shift, and activities of daily living.
Procedure: Respiratory rehabilitation — Forced expiration, forced inspiration (thoracal expansion exercise), coughing exercise, incentive spirometric trainer, diaphragmatic respiration exercise, autogenic drainage, percussion.
  Arms: Respiratory rehabilitation

SUMMARY:
This study evaluates the effects of respiratory exercises on respiratory function test parameters and ultrasonographic diaphragmatic measurements. Half of the hemiplegic patients will receive respiratory and neurophysiological exercises, while other half will receive only neurophysiological exercises.

DETAILED DESCRIPTION:
After stroke, diaphragm, the most important muscle of respiration, is wasted as well as the other muscles of the affected side.

Ultrasonography is a non-invasive, practical, low cost utility that may measure the thickness of diaphragm in maximum expiration and inspiration thus examining the functionality of the muscle. Correlation between respiratory functional tests and diaphragm ultrasonography has been proven in recent literature. In this manner, the aim of this study is twofold. First is to determine whether ultrasonography can be used practically to evaluate the respiratory functions of the patients after stroke. Respiratory function tests will be used for the correlation analysis. Second is to evaluate the effectiveness of respiratory exercises via diaphragm ultrasonography and respiratory function tests.

ELIGIBILITY:
Inclusion Criteria:

* Stroke confirmed radiologically
* Unilateral hemiplegia
* First stroke episode
* Mini Mental score ≥ 24

Exclusion Criteria:

* Unable to consent and understand
* Chronic cardiac disease
* Pulmonary disease (asthma, restrictive or obstructive pulmonary disease)
* Facial paralysis
* History of thoracic or abdominal surgery
* Being alcoholic
* Using psychotropic drugs

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2019-05-01 (Actual); Primary Completion 2020-02-01 (Actual); Study Completion 2020-02-01 (Actual)

PRIMARY OUTCOMES:
Forced vital capacity (FVC) | 6 weeks
  The amount of air that can be forcibly exhaled from the lungs after taking the deepest breath possible. Measured by spirometry. >80% is normal. If the value is lower than the normal limit it indicates either an obstructive or restrictive disease. The lower values show a poorer outcome
Forced expiratory volume in one second (FEV1) | 6 weeks
  The maximal amount of air you can forcefully exhale in one second. Measured by spirometry. >80% is normal. If there is an obstruction, this measurement shows the severity of the obstruciton. The lower values show a poorer outcome.
Tiffeneau-Pinelli index | 6 weeks
  A calculated ratio used in the diagnosis of obstructive and restrictive lung disease. Calculated as FEV1/FVC. >80% is normal. ≤80% indicates an obstructive pulmonary disease.
Forced expiratory flow at 25% and 75% (FEF 25-75%) | 6 weeks
  The average forced expiratory flow during the mid (25% - 75%) portion of the FVC. Shows small and medium airway obstruction. >70% is normal. It shows the small airways impariment
Diaphragmatic thickening fraction (TF) | 6 weeks
  Thickness of the diaphragm is measured from the zone of apposition (subcostal area between anterior axillary line and mid-axillary line) via ultrasonography. After diaphragm thickness in end expiration (thickness in functional residual capacity- TFRC) and in end inspiration (thickness in total lung capacity- TTLC) are obtained. Thickening fraction is calculated as [TTLC-TFRC/TFRC]x100. A higher value shows a better outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Ozan Volkan Yurdakul, MD, Study Director — Bezmialem University
Locations (1):
- Bezmialem Vakıf Univesity, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Jung KJ, Park JY, Hwang DW, Kim JH, Kim JH. Ultrasonographic diaphragmatic motion analysis and its correlation with pulmonary function in hemiplegic stroke patients. Ann Rehabil Med. 2014 Feb;38(1):29-37. doi: 10.5535/arm.2014.38.1.29. Epub 2014 Feb 25. PMID 24639923
- [Background] Kim M, Lee K, Cho J, Lee W. Diaphragm Thickness and Inspiratory Muscle Functions in Chronic Stroke Patients. Med Sci Monit. 2017 Mar 11;23:1247-1253. doi: 10.12659/msm.900529. PMID 28284044
- [Background] Cardenas LZ, Santana PV, Caruso P, Ribeiro de Carvalho CR, Pereira de Albuquerque AL. Diaphragmatic Ultrasound Correlates with Inspiratory Muscle Strength and Pulmonary Function in Healthy Subjects. Ultrasound Med Biol. 2018 Apr;44(4):786-793. doi: 10.1016/j.ultrasmedbio.2017.11.020. Epub 2018 Jan 17. PMID 29373153